CLINICAL TRIAL: NCT03338972
Title: A Phase I Study of Adoptive Immunotherapy for Advanced B-Cell Maturation Antigen (BCMA)+ Multiple Myeloma With Autologous CD4+ and CD8+ T Cells Engineered to Express a BCMA-Specific Chimeric Antigen Receptor
Brief Title: Immunotherapy With BCMA CAR-T Cells in Treating Patients With BCMA Positive Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Juno Therapeutics, Inc., a Bristol-Myers Squibb Company (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Damian Green, Associate Professor, Fred Hutchinson Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9762; NCI-2017-01932 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9762 (Other: Fred Hutch/University of Washington Cancer Consortium); RG9217023 (Other: Fred Hutch/University of Washington Cancer Consortium); P01CA018029 (NIH)
Record Dates: First submitted 2017-11-07; First posted 2017-11-09 (Actual); Results first posted 2022-08-05 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclophosphamide; fludarabine; Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment (chemotherapy, BCMA CAR-T cells) at dose level 1 (Experimental): Patients undergo leukapheresis. Patients then receive cyclophosphamide and fludarabine on days -4 to -2. Beginning to 36-96 days after chemotherapy, patients receive BCMA-specific CAR-expressing T lymphocytes IV over 20-30 minutes on day 0. Patients may receive a second dose of BCMA-specific CAR-expressing T lymphocytes IV with or without additional cytoreductive chemotherapy at the discretion of the principal investigator or their designee (sub-investigator).
  Arm 1 contains patients treated as dose level 1 (50 x 10^6 EGFRt cells)
  Interventions: Biological: Autologous Anti-BCMA-CAR-expressing CD4+/CD8+ T-lymphocytes FCARH143; Drug: Cyclophosphamide; Drug: Fludarabine; Procedure: Leukapheresis
- Treatment (chemotherapy, BCMA CAR-T cells) at dose level 2 (Experimental): Patients undergo leukapheresis. Patients then receive cyclophosphamide and fludarabine on days -4 to -2. Beginning to 36-96 days after chemotherapy, patients receive BCMA-specific CAR-expressing T lymphocytes IV over 20-30 minutes on day 0. Patients may receive a second dose of BCMA-specific CAR-expressing T lymphocytes IV with or without additional cytoreductive chemotherapy at the discretion of the principal investigator or their designee (sub-investigator).
  Arm 2 contains patients treated as dose level 2 (150 x 10^6 EGFRt cells)
  Interventions: Biological: Autologous Anti-BCMA-CAR-expressing CD4+/CD8+ T-lymphocytes FCARH143; Drug: Cyclophosphamide; Drug: Fludarabine; Procedure: Leukapheresis
- Treatment (chemotherapy, BCMA CAR-T cells) at dose level 3 (Experimental): Patients undergo leukapheresis. Patients then receive cyclophosphamide and fludarabine on days -4 to -2. Beginning to 36-96 days after chemotherapy, patients receive BCMA-specific CAR-expressing T lymphocytes IV over 20-30 minutes on day 0. Patients may receive a second dose of BCMA-specific CAR-expressing T lymphocytes IV with or without additional cytoreductive chemotherapy at the discretion of the principal investigator or their designee (sub-investigator).
  Arm 3 contains patients treated as dose level 3 (300 x 10^6 EGFRt cells)
  Interventions: Biological: Autologous Anti-BCMA-CAR-expressing CD4+/CD8+ T-lymphocytes FCARH143; Drug: Cyclophosphamide; Drug: Fludarabine; Procedure: Leukapheresis
- Treatment (chemotherapy, BCMA CAR-T cells) at dose level 4 (Experimental): Patients undergo leukapheresis. Patients then receive cyclophosphamide and fludarabine on days -4 to -2. Beginning to 36-96 days after chemotherapy, patients receive BCMA-specific CAR-expressing T lymphocytes IV over 20-30 minutes on day 0. Patients may receive a second dose of BCMA-specific CAR-expressing T lymphocytes IV with or without additional cytoreductive chemotherapy at the discretion of the principal investigator or their designee (sub-investigator).
  Arm 4 contains patients treated as dose level 4 (450 x 10^6 EGFRt cells)
  Interventions: Biological: Autologous Anti-BCMA-CAR-expressing CD4+/CD8+ T-lymphocytes FCARH143; Drug: Cyclophosphamide; Drug: Fludarabine; Procedure: Leukapheresis

INTERVENTIONS:
Biological: Autologous Anti-BCMA-CAR-expressing CD4+/CD8+ T-lymphocytes FCARH143 — Given IV
  Other Names: Autologous Anti-BCMA-CAR CD4+/CD8+ Cells; Autologous Anti-BCMA-CAR-expressing CD8+ and CD4+ T-lymphocytes; BCMA CAR-CD4+/CD8+ T-cells; BCMA-specific CAR-expressing CD4+/CD8+ T-lymphocytes; FCARH143
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocytopheresis; Therapeutic Leukopheresis

SUMMARY:
This phase I trial studies the side effects and best dose of BCMA CAR-T cells in treating patients with BCMA positive multiple myeloma that has come back or does not respond to treatment. T cells are a type of white blood cell and a major component of the immune system. T-cells that have been genetically modified in the laboratory express BCMA and may kill cancer cells with the protein BCMA on their surface. Giving chemotherapy before BCMA CAR-T cells may reduce the amount of disease and to cause a low lymphocyte (white blood cell) count in the blood, which may help the infused BCMA CAR-T cells survive and expand.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety of adoptive therapy with ex vivo expanded autologous CD8+ plus CD4+ T cells transduced to express a human B cell maturation antigen (BCMA)-targeting chimeric antigen receptor (CAR) for patients with relapsed or treatment refractory multiple myeloma.

SECONDARY OBJECTIVES:

I. To determine the duration of in vivo persistence and the phenotype of long lived CAR-T cells.

II. To determine the degree to which adoptively transferred T cells traffic to multiple myeloma (MM) cells in the bone marrow (BM) and function in vivo.

III. To estimate the antitumor activity of adoptively transferred BCMA-specific CAR-expressing T lymphocytes (BCMA CAR-T cells).

OUTLINE: This is a dose-escalation study of BCMA-specific CAR-expressing T lymphocytes.

Patients undergo leukapheresis to obtain their immune cells, from which CAR-T cells are produced. A few weeks later, patients then receive cyclophosphamide and fludarabine on days -4 to -2. Beginning 36-96 hours after chemotherapy, patients receive BCMA-specific CAR-expressing T lymphocytes intravenously (IV) over 20-30 minutes on day 0. Patients may receive a second dose of BCMA-specific CAR-expressing T lymphocytes IV with or without additional cytoreductive chemotherapy at the discretion of the principal investigator or their designee (sub-investigator).

After completion of study treatment, patients are followed up at 60, 90, 120, 180, and 365 days and then annually up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Have the capacity to give informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status score =< 2.
* Have measurable disease by International Myeloma Working Group (IMWG) criteria based on one or more of the following findings:

  * Serum M-protein >= 1 g/dL
  * Urine M-protein >= 200 mg/24 hour
  * Involved serum free light chain (sFLC) level >= 10 mg/dL with abnormal kappa/lambda ratio
  * Measurable biopsy-proven plasmacytomas (>= 1 lesion that has a single diameter >= 2 cm)
  * Bone marrow plasma cells >= 30%
* Have a diagnosis of BCMA+ MM (>= 5% BCMA+ by flow cytometry on CD138 co-expressing plasma cells obtained within 45 days of study enrollment); the MM diagnosis must be confirmed by internal pathology review of a fresh biopsy specimen at the Fred Hutchinson Cancer Research Center (FHCRC)/Seattle Cancer Care Alliance (SCCA)
* Have relapsed or treatment refractory disease with >= 10% CD138+ malignant plasma cells (IHC) on BM core biopsy, either:

  * Following autologous stem cell transplant (ASCT)
  * Or, if a patient has not yet undergone ASCT, the individual must:

    * Be transplant ineligible, due to age, comorbidity, patient choice, insurance reasons, concerns of rapidly progressive disease, and/or discretion of attending physician and principal investigator and,
    * Demonstrate disease that persists after > 4 cycles of induction therapy and that is double refractory (persistence/progression) after therapy with both a proteasome inhibitor and immunomodulatory drug (IMiD) administered either in tandem, or in sequence; > 4 cycles of therapy are not required for patients with a diagnosis of plasma cell leukemia

      * Patients receiving retreatment do not need to meet the > 10% CD138+ malignant plasma cells (immunohistochemistry staining method [IHC]) on BM core biopsy
* Male and female patients of reproductive potential must be willing to use an effect contraceptive method before, during, and for at least 4 months after the CAR T cell infusion

Exclusion Criteria:

* History of another primary malignancy that requires intervention beyond surveillance or that has not been in remission for at least 1 year (the following are exempt from the 1 year limit: non-melanoma skin cancer, curatively treated localized prostate cancer, and cervical carcinoma in situ on biopsy or a squamous intraepithelial lesion on papanicolaou [PAP] smear)
* Active hepatitis B, hepatitis C at the time of screening
* Patients who are (human immunodeficiency virus [HIV]) seropositive
* Subjects with uncontrolled active infection
* > 1 hospital admission (lasting 5 days or more) for documented infection in prior 6 months
* Presence of acute or chronic graft-versus-host disease (GVHD) requiring active treatment unless limited to skin involvement and managed with topical steroid therapy alone
* History of any one of the following cardiovascular conditions within the past 6 months: Class III or IV heart failure as defined by the New York Heart Association (NYHA), cardiac angioplasty or stenting, myocardial infarction, unstable angina, or other clinically significant cardiac disease as determined by the principal investigator (PI) or designee
* History of clinically relevant or active central nervous system (CNS) pathology such as epilepsy, seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis, active central nervous system MM involvement and/or carcinomatous meningitis; subjects with previously treated central nervous systems involvement may participate, provided they are free of disease in the CNS (documented by flow cytometry performed on the cerebrospinal fluid [CSF] within 14 days of enrollment) and have no evidence of new sites of CNS activity
* Pregnant or breastfeeding females
* Allogeneic HSCT or donor lymphocyte infusion within 90 days of leukapheresis.
* Use of any of the following:

  * Therapeutic doses of corticosteroids (defined as > 20 mg/day prednisone or equivalent) within 7 days prior to leukapheresis; physiologic replacement, topical, and inhaled steroids are permitted
  * Cytotoxic chemotherapeutic agents within 1 week of leukapheresis; oral chemotherapeutic agents are allowed if at least 3 half-lives have elapsed prior to leukapheresis
  * Lymphotoxic chemotherapeutic agents within 2 weeks of leukapheresis
  * Daratumumab (or other anti-CD38 therapy) within 30 days of leukapheresis
  * Experimental agents within 4 weeks of leukapheresis unless progression is documented on therapy and at least 3 half-lives have elapsed prior to leukapheresis
* Absolute neutrophil count (ANC) < 1000/mm^3, or per PI discretion if cytopenia thought to be related to underlying myeloma.
* Hemoglobin (Hgb) < 8 mg/dl, or per PI discretion if cytopenia thought to be related to underlying myeloma.
* Platelet count < 50,000/mm^3, or per PI discretion if cytopenia thought to be related to underlying myeloma.
* Active autoimmune disease requiring immunosuppressive therapy
* Major organ dysfunction defined as:

  * Creatinine clearance < 20 ml/min
  * Significant hepatic dysfunction (serum glutamic-oxaloacetic transaminase [SGOT] > 5 x upper limit of normal; bilirubin > 3.0 mg/dL)
  * Forced expiratory volume in 1 second (FEV1) of < 50% predicted or diffusion capacity of the lung for carbon monoxide (DLCO) (corrected) < 40% (patients with clinically significant pulmonary dysfunction, as determined by medical history and physical exam should undergo pulmonary function testing)
* Anticipated survival of < 3 months
* Contraindication to cyclophosphamide or fludarabine chemotherapy
* Patients with known AL subtype amyloidosis
* Uncontrolled medical, psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol, as judged by the PI; or unwillingness or inability to follow the procedures required in the protocol

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2022-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Damian J. Green, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Tuazon SA, Portuguese AJ, Pont MJ, Cowan AJ, Cole GO, Sather BD, Song X, Thomas S, Wood BL, Blake M, Works MG, Shadman M, Liang EC, Wu QV, Voutsinas JM, Gooley TA, Turtle CJ, Till BG, Coffey DG, Maloney DG, Riddell SR, Green DJ. A phase 1 trial of fully human BCMA CAR-T therapy for relapsed/refractory multiple myeloma with 5-year follow-up. Blood. 2025 Jul 31;146(5):535-545. doi: 10.1182/blood.2024027681. PMID 40198877

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3 patients withdrew consent after enrollment and did not move on to treatment. These 3 patients were not assigned to a dose level.
Groups:
- Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 1: Patients undergo leukapheresis. Patients then receive cyclophosphamide and fludarabine on days -4 to -2. Beginning to 36-96 days after chemotherapy, patients receive BCMA-specific CAR-expressing T lymphocytes IV over 20-30 minutes on day 0. Patients may receive a second dose of BCMA-specific CAR-expressing T lymphocytes IV with or without additional cytoreductive chemotherapy at the discretion of the principal investigator or their designee (sub-investigator).
  Arm 1 contains patients treated as dose level 1 (50 x 10^6 EGFRt cells)
  Autologous Anti-BCMA-CAR-expressing CD4+/CD8+ T-lymphocytes FCARH143: Given IV
  Cyclophosphamide: Given IV
  Fludarabine: Given IV
  Leukapheresis: Undergo leukapheresis
- Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 2: Patients undergo leukapheresis. Patients then receive cyclophosphamide and fludarabine on days -4 to -2. Beginning to 36-96 days after chemotherapy, patients receive BCMA-specific CAR-expressing T lymphocytes IV over 20-30 minutes on day 0. Patients may receive a second dose of BCMA-specific CAR-expressing T lymphocytes IV with or without additional cytoreductive chemotherapy at the discretion of the principal investigator or their designee (sub-investigator).
  Arm 2 contains patients treated as dose level 2 (150 x 10^6 EGFRt cells)
  Autologous Anti-BCMA-CAR-expressing CD4+/CD8+ T-lymphocytes FCARH143: Given IV
  Cyclophosphamide: Given IV
  Fludarabine: Given IV
  Leukapheresis: Undergo leukapheresis
- Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 3: Patients undergo leukapheresis. Patients then receive cyclophosphamide and fludarabine on days -4 to -2. Beginning to 36-96 days after chemotherapy, patients receive BCMA-specific CAR-expressing T lymphocytes IV over 20-30 minutes on day 0. Patients may receive a second dose of BCMA-specific CAR-expressing T lymphocytes IV with or without additional cytoreductive chemotherapy at the discretion of the principal investigator or their designee (sub-investigator).
  Arm 3 contains patients treated as dose level 3 (300 x 10^6 EGFRt cells)
  Autologous Anti-BCMA-CAR-expressing CD4+/CD8+ T-lymphocytes FCARH143: Given IV
  Cyclophosphamide: Given IV
  Fludarabine: Given IV
  Leukapheresis: Undergo leukapheresis
- Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 4: Patients undergo leukapheresis. Patients then receive cyclophosphamide and fludarabine on days -4 to -2. Beginning to 36-96 days after chemotherapy, patients receive BCMA-specific CAR-expressing T lymphocytes IV over 20-30 minutes on day 0. Patients may receive a second dose of BCMA-specific CAR-expressing T lymphocytes IV with or without additional cytoreductive chemotherapy at the discretion of the principal investigator or their designee (sub-investigator).
  Arm 4 contains patients treated as dose level 4 (450 x 10^6 EGFRt cells)
  Autologous Anti-BCMA-CAR-expressing CD4+/CD8+ T-lymphocytes FCARH143: Given IV
  Cyclophosphamide: Given IV
  Fludarabine: Given IV
  Leukapheresis: Undergo leukapheresis
Period: Overall Study
Arm/Group | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 1 | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 2 | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 3 | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 4
Started | 7 | 8 | 7 | 3
Completed | 5 | 7 | 7 | 3
Not Completed | 2 | 1 | 0 | 0
Not completed — Death | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 1 | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 2 | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 3 | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 4 | Total
Number analyzed (Participants) | 7 | 8 | 7 | 3 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 5 | 1 | 14
  >=65 years | 3 | 4 | 2 | 2 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 3 | 1 | 9
  Male | 5 | 5 | 4 | 2 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 6 | 8 | 7 | 2 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 6 | 7 | 6 | 2 | 21
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 7 | 3 | 25

OUTCOME MEASURES:

1. Primary Outcome: Dose-limiting Toxicities (DLT) Rate
Description: Observed DLT rates will be summarized based on the DLT-Evaluable analysis set. Outcome will be reported as count of participants in each arm who experienced a DLT. No patients received more than one CAR T cell infusion, so DLT assessment period was only 28 days after first and only CAR T infusion for all patients.
Time Frame: Up to 28 days after CAR T cell infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 1 | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 2 | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 3 | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 4
Number analyzed (Participants) | 7 | 8 | 7 | 3
Participants | 0 | 0 | 1 | 0

2. Primary Outcome: Count of Patients That Experienced Adverse Events
Description: Toxicity graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 No patients received more than one CAR T cell infusion, so AE assessment period was only 28 days after first and only CAR T infusion for all patients.
Time Frame: Up to 28 days after CAR T-cell infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 1 | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 2 | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 3 | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 4
Number analyzed (Participants) | 7 | 8 | 7 | 3
Participants | 7 | 8 | 7 | 3

3. Secondary Outcome: Duration of Persistence of Adoptively Transferred BCMA CAR-T Cells
Description: Persistence of CART cells is tested by qPCR in PBMC.
Time Frame: Assessed from Baseline up to a maximum of 537 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 1 | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 2 | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 3 | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 4
Number analyzed (Participants) | 7 | 8 | 7 | 3
Days | 134 [104 to 182] | 110 [64 to 169] | 386 [282 to 537] | 236 [133 to 309]

4. Secondary Outcome: Number of Participants With Detectable BCMA CART Cell Migration to Primary Disease Site (Bone Marrow) at Day 28
Time Frame: Baseline up to Day 28
Population: CART cell migration to bone marrow was identified in all patients for whom a Day 28 bone marrow biopsy specimen was available (19 out of 19). In 6 cases, biopsy was not performed due to patient clinical status or bone marrow biopsy was attempted but no aspirate could be collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 1 | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 2 | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 3 | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 4
Number analyzed (Participants) | 5 | 7 | 5 | 2
Participants | 5 | 7 | 5 | 2

5. Secondary Outcome: Objective Response Rate (ORR)
Description: Number of patients with a best response of either complete response, stringent complete response, very good partial response or partial response, assessed using modified International Myeloma Working group response criteria.
Time Frame: Baseline up to 3 months after CART infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 1 | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 2 | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 3 | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 4
Number analyzed (Participants) | 7 | 8 | 7 | 3
Participants | 7 | 8 | 7 | 3

6. Secondary Outcome: Progression-free Survival (PFS)
Description: Outcome is reported as the count of participants who were alive at the 1 year post treatment mark and did not experience disease progression by the 1 year post treatment mark.
Time Frame: Assessed up to 1 year after CART infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 1 | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 2 | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 3 | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 4
Number analyzed (Participants) | 7 | 8 | 7 | 3
Participants | 3 | 5 | 5 | 2

7. Secondary Outcome: Overall Survival (OS)
Description: Outcome is reported as a count of participants who were alive at the 1 year post-infusion timepoint.
Time Frame: Assessed up to 1 year after CART infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 1 | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 2 | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 3 | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 4
Number analyzed (Participants) | 7 | 8 | 7 | 3
Participants | 3 | 5 | 7 | 3

ADVERSE EVENTS:
Time Frame: Adverse Events were assessed up to 28 days after CAR T-cell infusion. No patients received more than one CAR T cell infusion, so AE assessment period was only 28 days after first and only CAR T infusion for all patients. All-Cause Mortality was assessed up to 1 year.
Description: An Adverse Event (AE) is any undesirable experience associated with the use of a medical product in a patient. The NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.
Arm/Group | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 1 | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 2 | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 3 | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 4
All-Cause Mortality (participants affected / at risk) | 4/7 | 3/8 | 0/7 | 0/3
Serious Adverse Events (participants affected / at risk) | 5/7 | 8/8 | 5/7 | 3/3
Other Adverse Events (participants affected / at risk) | 7/7 | 8/8 | 7/7 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 1 (N=7) | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 2 (N=8) | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 3 (N=7) | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 4 (N=3)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 3 (3) | 3 (5) | 1 (1) | 1 (1)
NEUTROPENIC FEVER (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FEVER (General disorders) | 2 (4) | 5 (5) | 3 (4) | 1 (1)
CYTOKINE RELEASE SYNDROME (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INFECTIONS AND INFESTATIONS - OTHER, LYSINIBACILLUS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LUNG INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 1 (N=7) | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 2 (N=8) | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 3 (N=7) | Treatment (Chemotherapy, BCMA CAR-T Cells) at Dose Level 4 (N=3)
ANEMIA (Blood and lymphatic system disorders) | 5 (19) | 8 (19) | 5 (12) | 2 (5)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 3 (5) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 2 (2) | 2 (3) | 2 (4) | 0 (0)
FEVER (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PAIN (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PAIN NOS (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
CYTOKINE RELEASE SYNDROME (Immune system disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
INFECTIONS AND INFESTATIONS - OTHER, CMV (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY : BACTEREMIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ALANINE AMINOTRASFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
BILIRUBIN INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CARDIAC TROPONIN INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
LYMPHOCYTE COUNT DECREASED (Investigations) | 7 (19) | 8 (23) | 7 (32) | 3 (7)
NEUTROPHIL COUNT DECREASE (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 7 (19) | 8 (20) | 6 (22) | 3 (9)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
PLATELET COUNT DECREASED (Investigations) | 6 (11) | 5 (10) | 4 (25) | 3 (9)
WHITE BLOOD CELL DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
WHITE BLOOD CELL DECREASED (Investigations) | 7 (15) | 8 (18) | 7 (24) | 3 (11)
ANOREXIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERKALEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERURICEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (4) | 0 (0)
HYPOKALEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
HYPONATREMIA (Metabolism and nutrition disorders) | 2 (3) | 1 (2) | 3 (6) | 1 (1)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 2 (3) | 5 (5) | 2 (3) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (4) | 0 (0)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BONE PAIN (RIB) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
HIP PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PAIN R HIP (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COGNITIVE DISTURBANCE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSPHASIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (7) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
MUSCLE WEAKNESS LEFT-SIDED (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NERVOUS SYSTEM DISORDERS - OTHER, SPECIFY - LEFT SIDE NEGLIGENCE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONFUSION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
PROTEINURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 4 (4) | 0 (0)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 1 (2) | 2 (2) | 3 (7) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1) | 1 (1) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT03338972/Prot_SAP_000.pdf